CLINICAL TRIAL: NCT04876976
Title: Isoamyl 2-Cyanoacrylate Interposition in the Urethro-cutaneous Fistula Repair: A Randomized Controlled Trial.
Brief Title: Isoamyl 2-Cyanoacrylate in the Urethro-cutaneous Fistula Repair
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Maher Gamil Ahmed Higazy, assistant lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS 75/2018
Record Dates: First submitted 2021-04-29; First posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Hypospadias
Keywords: Isoamyl 2-cyanoacrylate; urethrocutaneous fistula; fistula repair; hypospadias
MeSH Terms: conditions — Hypospadias | interventions — Bucrylate

STUDY DESIGN:
Intervention Model Description: Cases of group (I) underwent multilayered closure using dartos facial flap and cyanoacrylate glue as an interposition layer.
  Cases of the control group (II) underwent the same procedure without using cyanoacrylate.
Who Masked: Participant
Masking Description: patients and their relatives were blinded to the type of the intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cases of group (I) cyanoacrylate glue (Experimental): Cases of group (I) underwent multilayered closure using dartos facial flap and cyanoacrylate glue as an interposition layer.
  Interventions: Drug: Cyanoacrylate, Isobutyl
- Cases of the control group (II) , classic repair (Active Comparator): Cases of the control group (II) underwent the same procedure without using cyanoacrylate.
  Interventions: Procedure: Classic surgical repair

INTERVENTIONS:
Drug: Cyanoacrylate, Isobutyl — using cyanoacrylate in the surgical repair of urethro-cutaneous fistula
  Arms: Cases of group (I) cyanoacrylate glue
Procedure: Classic surgical repair — classical repair of urethro-cutaneous fistula without the use of cyanoacryalte
  Arms: Cases of the control group (II) , classic repair

SUMMARY:
cyanoacrylate has an impact that may aid in the successful repair of urethra-cutaneous fistula (UCF) that occur after hypospadias surgical repair

DETAILED DESCRIPTION:
Hypospadias is a common congenital urological birth defect. Urethro-cutaneous fistula (UCF) is the most common complication of surgical repair hypospadias and it remains the primary concern of surgeons dealing with hypospadias repair.

cyanoacrylate has been reported to enhance the healing process. this study tries to evaluate the clinical impact of cyanoacrylate on the repair of urethro-cutaneous fistula after surgical repair of hypospadias

this study evaluates the impact of using cyanoacrylate as an interposition substance in surgical repair of UCF after hypospadias in comparison to the classic surgical repair technique

ELIGIBILITY:
Inclusion Criteria:

* Patients with Urethro-cutaneous fistula regardless of their age were included in our study.

Exclusion Criteria:

* Patients with fistula size more than 5 mm
* multiple fistulas
* uncorrected obstruction distal to the fistula
* necrotic tissue
* active infection at the fistula site
* severely scarred skin
* deficient dartos around the fistula
* fistulas more proximal to the mid penile position
* recurrent fistulas
* previous history of hypersensitivity to cyanoacrylate-based products

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Hypospadias is a male urethral congenital anomaly
Enrollment: 40 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
successful repair of the fistula | 6 months after surgery
  surgical outcome regarding the repair of urethro-cutaneous fistula, whether adequate healing occurred or recurrence is present

SECONDARY OUTCOMES:
postoperative complications | 6 months after surgery
  report of the possible postoperative complications of both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Urology department - ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided